CLINICAL TRIAL: NCT03362307
Title: Use Low-Level Laser and Light-Emitting Diodes in Dental Implants
Brief Title: Can Combination of Low-Level Laser and Light-Emitting Diodes Enhance Stability of Dental Implants?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Collaborators: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Reza Tabrizi, associate Professor, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Fr1396
Record Dates: First submitted 2017-11-28; First posted 2017-12-05 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Dental Implant Healing
Keywords: Low-Level Light Therapy, Osseointegration

STUDY DESIGN:
Intervention Model Description: Subjects were aligned based on computer randomization in two groups: In group 1(intervention), subjects received LLL and LED after implant placement and in group 2 (control) the same device was used while device was off.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser Emitting group (Active Comparator): subjects received Low-Level Laser and Light-Emitting Diodes after implant placement
  Interventions: Device: Low-Level Laser and Light-Emitting Diodes; Device: Dental implant placement
- Non Emitting group (Placebo Comparator): In laser emitiiing group, subjects received Low-Level Laser and Light-Emitting Diodes after implant placement and in Non-emitting group,the same device was used while device was off.
  Interventions: Device: Low-Level Laser and Light-Emitting Diodes; Device: Dental implant placement

INTERVENTIONS:
Device: Low-Level Laser and Light-Emitting Diodes — Combination of Low-Level Laser and Light-Emitting Diodes were used after dental implant placement for enhancement of stability
Device: Dental implant placement — A dental implant with 4.8X 10 mm (Zimmer, USA) size was placed at the posterior of the mandible

SUMMARY:
Subjects were assigned in two groups: In group 1, subjects received LLL and LED 20 min/day for 10 days after implant insertion, subjects in group 2did not undergo LLL and LED. implant stability quotients(ISQs) were measured in 0,10,21,42 and 63 days after implant placement.

DETAILED DESCRIPTION:
Subjects eligible for study inclusion had an edentulous area at the first molar of the mandible and needed a dental implant. Subjects were excluded from study enrollment if they had any diseases that affect bone, smoking, insufficient bone in the edentulous area which needs bone augmentation, failed to return for follow-up, or refused study enrollment.

All implants were placed at least 3 months after tooth removal. The size of implants was 4.8X 10 mm (Zimmer, USA) Subjects were aligned based on computer randomization in two groups: In group 1(intervention), subjects received LLL and LED after implant placement and in group 2 (control) the same device was used while device was off.

A portable device was applied for irradiation of the intervention group with combination of 810nm laser and 632nm LED.

Subjects in group 1 underwent LLL 15 mw/cm2 and LED 10 mw/cm2 20 min every day for 10 days.

The mesiodistal and buccolingual directions were measured and the mean implant stability quotients (ISQs) were determined. The RFA measurements were performed in immediate after insertion (time0) 10 days (time1), 3 weeks (time2), 6 weeks(time3) and 9(time 4) weeks after implant placement.

ELIGIBILITY:
Inclusion Criteria:

* subjects eligible for study inclusion had an edentulous area at the first molar of the mandible and needed a dental implant

Exclusion Criteria:

* . Subjects were excluded from study enrollment if they had any diseases that affect bone, smoking, insufficient bone in the edentulous area which needs bone augmentation, failed to return for follow-up, or refused study enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2015-01-01 (Actual); Study Completion 2015-09-30 (Actual)

PRIMARY OUTCOMES:
Resonance frequency analysis | Immidate after implant placement (time 0)
  The stability of the implants was evaluated with resonance frequency analysis by the Osstell device
Resonance frequency analysis | 10 days (time1) after implant placement
  The stability of the implants was evaluated with resonance frequency analysis by the Osstell device
Resonance frequency analysis | Three weeks after implant placement (time 2)
  The stability of the implants was evaluated with resonance frequency analysis by the Osstell device
Resonance frequency analysis | Six weeks after implant placement (time 3)
  The stability of the implants was evaluated with resonance frequency analysis by the Osstell device
Resonance frequency analysis | Nine weeks after implant placement(time 4)
  The stability of the implants was evaluated with resonance frequency analysis by the Osstell device

IPD SHARING:
Plan to Share IPD: Undecided